CLINICAL TRIAL: NCT02341755
Title: Dual Energy Computerized Tomography (DE-CT) for Evaluation of Obstructive Intestinallesions in Patients With Crohn's Disease
Brief Title: Dual Energy Computerized Tomography (DE-CT) in Patients With Crohn's Disease
Status: Terminated | Type: Observational
Why Stopped: Interim analysis was sufficient to demonstrate accuracy of the evaluated test
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Tomer Adar, Senior physician in internal medicine, senior gastroenterologist, Shaare Zedek Medical Center
Other Study IDs: 47/12
Record Dates: First submitted 2015-01-11; First posted 2015-01-19 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to evaluate the accuracy of dual energy computerized tomography (DE-CT) in predicting the need for surgery in patients with Crohn's disease and intestinal lesions with obstructive symptoms.

Patients with known Crohn's disease which were scheduled to perform abdominal CT for obstructive symptoms preformed it in a dual energy protocol and then followed for an outcome of surgery. DE-CT parameters were then compared between patients who underwent surgery and those who did not.

DETAILED DESCRIPTION:
INTRODUCTION Intestinal strictures are common in patients with Crohn's (CD) disease and may result in intestinal obstruction. Current available imaging studies can usually identify and locate the stricture, but can not reliably differentiate the patients who will require surgery from those who will respond to medical therapy.

Dual Energy computerized tomography (DE-CT) uses two energy sources using high and low tube voltage, thus creating two data sets. Dedicated software creates overlay of the low and high energy images, in which enhancement of tissues with iodine can be better appreciated and quantified compared to standard CT. The investigators hypothesize that dual energy can better visualize the iodine uptake in bowl wall as a marker of inflammation within intestinal lesions, and may help in identifying the patients who will or will not require surgery.

AIM To evaluate the efficacy of DE-CT studies in predicting need for surgery within 3 months.

METHODS Patients with known CD undergoing abdominal CT for possible obstructive presentation prospectively underwent a DE-CT using intravenous iodinated contrast material, and were followed for 3 months for an outcome of surgery.

The DE-CT was interpreted by a radiologist blinded to the clinical outcome, and the attending physicians of the patients were blinded to the interpretation of the DE-CT. DE-CT parameters were then compared between patients who underwent surgery and those who did not. Receiver operating characteristic (ROC) curve analysis was used to find the optimal cut off point to distinguish between patients which did or did not eventually underwent surgery. Based on the cut off points found from the ROC analysis, the negative and positive predictive values were calculated.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years,
* known Crohn's disease (at least 3 moths prior)
* obstructive symptoms
* scheduled for abdominal CT for evaluation of symptoms (regardless of participation in the study)

Exclusion Criteria:

* Pregnancy
* Contraindication to perform CT with IV contrast media

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known Crohn's disease undergoing abdominal CT for possible obstructive presentation
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2012-05; Primary Completion 2014-04 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Abdominal surgery | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Tomer Adar, MD, Principal Investigator — Shaare Zedek Medical Center affiliated with Hebrew University, Jerusalem, Israel.
Locations (1):
- Shaare Zedek Medical Center affiliated with Hebrew University, Jerusalem, Israel